CLINICAL TRIAL: NCT07302841
Title: A Clinical Study Evaluating the Efficacy and Safety of Tunlametinib in Combination With Chemotherapy and Cetuximab β in Patients With Advanced Pancreatic Cancer
Brief Title: Tunlametinib + AG + Cetuximab β as First-Line Therapy for Advanced Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-085-ST-005
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Cancer Non-resectable
Keywords: first-line therapy in treatment; MEK inhibitor; AG; Tunlametinib; Cetuximab β

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tunlametinib+gemcitabine+albumin paclitaxel + cetuximab β (Experimental)
  Interventions: Drug: Experimental: Tunlametinib+gemcitabine+albumin paclitaxel + cetuximab β

INTERVENTIONS:
Drug: Experimental: Tunlametinib+gemcitabine+albumin paclitaxel + cetuximab β — Tunlametinib + Gemcitabine + Albumin Paclitaxel + Cetuximab β. The dosage of Tunlametinib capsules is 9 mg, taken orally twice a day (BID), continuously administered; the dosage of Gemcitabine is 1000 mg/m2, intravenous infusion for more than 30 minutes, on days 1 and 8; Albumin Paclitaxel, 125 mg/m2, intravenous infusion, on days 1 and 8, with a cycle every 3 weeks; Cetuximab β: 500 mg/m², intravenous infusion, on day 1, with the injection duration exceeding 2 hours but not more than 4 hours, administered once every 2 weeks.

SUMMARY:
This study is a prospective, open-label, single-arm clinical trial evaluating the safety and efficacy of tunlametinib in combination with gemcitabine/albumin-bound paclitaxel and an EGFR monoclonal antibody as first-line therapy in treatment-naive subjects with advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Signing of a written informed consent form prior to enrolment;
2. Age > 18 years, males and females eligible;
3. Patients with histologically or pathologically confirmed advanced pancreatic cancer;
4. No prior systemic therapy;
5. At least one measurable lesion according to RECIST v1.1 assessment;
6. ECOG Performance Status: 0-1;
7. Expected survival greater than 12 weeks;
8. Major organ function meeting the following requirements:

   * Haemogram: Neutrophils ≥ 1.5 × 10⁹/L; Platelet count ≥ 100 × 10⁹/L; Haemoglobin ≥ 90 g/L; Maintenance of these haematological parameters without G-CSF, platelet transfusion, TPO infusion, blood transfusion, or erythropoietin support for 14 days prior to first dose.
   * Hepatic and Renal Function: Serum creatinine (SCr) ≤ 1.5 times the upper limit of normal (ULN) or creatinine clearance ≥ 50 ml/min (Cockcroft-Gault formula); Total bilirubin (TBIL) ≤ 3 times the upper limit of normal (ULN); Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels ≤ 5 times ULN; Urine protein <2+; if urine protein ≥2+, 24-hour urine protein quantification must show protein ≤1g;
   * Creatine kinase (CK) ≤ 1.5 × ULN
9. Normal coagulation function with no active bleeding or thrombotic disorders: International Normalised Ratio (INR) ≤ 1.5 × ULN; Activated Partial Thromboplastin Time (APTT) ≤ 1.5 × ULN; Prothrombin Time (PT) ≤ 1.5 × ULN;
10. Non-surgically sterilised or female patients of childbearing potential must use one medically approved contraceptive method (e.g., intrauterine device, oral contraceptive, condom) during study treatment and for 3 months post-treatment. Non-surgically sterilised female patients of childbearing potential must have negative serum or urinary hCG tests within 7 days prior to study entry and must not be lactating. Male subjects who are not surgically sterilised or who are of reproductive age must agree to use one medically approved contraceptive method with their partner during the study treatment period and for 3 months after the study treatment period.
11. Able to take oral medication;
12. The subject voluntarily participates in this study, demonstrates good compliance, and cooperates with safety and survival follow-up.

Exclusion Criteria:

1. Known contraindications affecting the investigator's choice of therapeutic agent (as per the latest prescribing information)
2. Receipt of any other investigational treatment within 4 weeks prior to study dosing initiation;
3. Undergoing major surgery (excluding biopsy, minor outpatient procedures such as vascular access placement) or experiencing severe trauma within 4 weeks prior to first dosing, or having scheduled major surgery within 30 days after first dosing (as determined by the investigator);
4. Previous receipt of anti-EGFR monoclonal antibodies, EGFR tyrosine kinase inhibitors, or other EGFR-targeted therapies (e.g., cetuximab, nintedanib, panitumumab);
5. Presence of clinically symptomatic third-space effusions uncontrollable by drainage or other methods (e.g., massive pleural effusion or ascites);
6. Symptomatic or untreated brain metastases, leptomeningeal metastases, or spinal cord compression, except for asymptomatic brain metastases (i.e., no progressive CNS symptoms attributable to brain lesions, no requirement for corticosteroids or antiepileptic drugs, and imaging confirmation of stable disease for ≥4 weeks); Patients undergoing stereotactic brain radiotherapy or surgery may be eligible if no disease progression is observed in the brain over a period of ≥3 months;
7. Cardiac impairment or clinically significant cardiovascular disease with uncontrolled cardiac symptoms or conditions, such as: (1) NYHA Class II or higher heart failure; (2) unstable angina pectoris; (3) myocardial infarction within the past year; (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention;
8. History or presence at screening of retinal disease, including: retinal vein occlusion (RVO), retinal artery occlusion, retinal vasculitis, diabetic retinopathy, hypertensive retinopathy, retinal capillaropathy (Costs disease), retinal pigment epithelial detachment (RPED); Presence of RVO risk factors at screening (e.g., uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulable syndromes); retinal diseases such as RPED;
9. Patients with interstitial lung disease or interstitial pneumonia, including clinically significant radiation pneumonitis (i.e., affecting activities of daily living or requiring intervention);
10. Known active pulmonary tuberculosis (TB); subjects suspected of active TB must undergo clinical evaluation to rule it out; known active syphilis infection;
11. Human immunodeficiency virus (HIV) antibody positive, syphilis antibody (Anti-TP) positive, hepatitis C virus (HCV) antibody positive with HCV RNA positive, hepatitis B virus surface antigen (HBsAg) positive with HBV DNA positive (HBsAg positive requires further testing for HBV DNA, HBV DNA ≥ 200 IU/ml, or ≥ 10³ copies/ml);
12. History of chronic inflammatory bowel disease or Crohn's disease requiring medical intervention (immunomodulators or surgery) within 12 months prior to treatment initiation;
13. Known history of acute or chronic pancreatitis within 6 months prior to study treatment initiation;
14. History of allogeneic bone marrow transplantation or organ transplantation;
15. Uncontrolled active infectious disease requiring intravenous antibiotics, antifungals, or antivirals within 2 weeks prior to first dosing, or unexplained fever >38.5°C during screening/prior to first dosing;
16. Uncorrectable electrolyte abnormalities (hypokalaemia, hypomagnesaemia, hypocalcaemia confirmed by blood biochemistry);
17. Past or current neuromuscular disorders associated with elevated CK levels (e.g., inflammatory myopathies, muscular dystrophies, amyotrophic lateral sclerosis, spinal muscular atrophy, rhabdomyolysis syndrome);
18. Arterial or venous thromboembolic events occurring within 6 months prior to first administration, such as cerebrovascular accidents (including transient ischaemic attacks, cerebral haemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
19. Presence of oesophageal or gastric varices, severe ulcers, unhealed wounds, gastrointestinal perforation, abdominal fistula, intra-abdominal abscess, or history of acute gastrointestinal haemorrhage within 6 months prior to first administration; occurrence of hypertensive crisis or hypertensive encephalopathy within 6 months prior to first administration; acute exacerbation of chronic obstructive pulmonary disease within 1 month prior to first administration;
20. Grade 3 bleeding events as defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v5.0) within 4 weeks prior to first dosing;
21. History of severe bleeding tendency or coagulation disorders; screening imaging demonstrating tumour encasement of major vessels or significant necrosis/cavitation, where the investigator deems participation may pose a bleeding risk;
22. Current radiographic or clinical evidence of significant gastrointestinal obstruction;
23. History of other malignancies within the past 5 years, except for patients with completely cured basal cell carcinoma or squamous cell carcinoma of the skin, cervical carcinoma in situ, and/or any malignancy that has been cured with no evidence of disease or at least 5 years of continuous disease-free status;
24. Known allergy to any component of the study drug;
25. History of defined neurological or psychiatric disorders, including epilepsy and dementia;
26. Failure of all relevant antineoplastic treatment toxicities to recover to Grade ≤1 (as assessed per NCI CTCAE V5.0) prior to study drug administration;
27. Concurrent use of other antineoplastic agents for concomitant therapy (bisphosphonates for bone metastases are acceptable);
28. Uncontrolled concomitant conditions, including but not limited to severe diabetes mellitus (fasting blood glucose > 250 mg/dl or 13.9 mmol/L) or other serious illnesses requiring systemic treatment;
29. Recipient of live or attenuated vaccines within 4 weeks prior to first dosing (Note: If enrolled, subjects must not receive live vaccines during study treatment or within 30 days after the last study drug dose);
30. Positive pregnancy test results in premenopausal female subjects (postmenopausal female subjects must have been amenorrheic for at least 12 months to be considered non-fertile); subjects of reproductive age (including female partners of male subjects) who are likely to become pregnant, are breastfeeding, or are unwilling to use effective contraception during the study period and for at least 30 days after the last dose of study medication;
31. Patients currently receiving intravenous or oral medications that are prohibited by the protocol due to their effects on CYP isoenzymes (strong inducers or inhibitors of CYP2C9 and CYP3A4) and cannot be discontinued at least one week prior to study treatment initiation and throughout the study period; patients taking narrow therapeutic index medications metabolised via CYP1A2;
32. Inability to swallow capsules, or refractory nausea and vomiting, malabsorption, extrahepatic bile diversion, or significant small bowel resection that may impair adequate absorption of the study drug;
33. Other circumstances deemed unsuitable for inclusion by the investigator. For example, family or social factors that may compromise the subject's safety or the collection of data and samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-06-20 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
ORR | 2 years

SECONDARY OUTCOMES:
PFS | 2 years
DCR | 2 years
DOR | 2 years
AEs | 2 years
OS | 2 years